CLINICAL TRIAL: NCT00032513
Title: Genetic Studies of Chronic Active Epstein-Barr Virus Infection
Brief Title: Genetic Studies of Chronic Active Epstein-Barr Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020147; 02-I-0147
Record Dates: First submitted 2002-03-22; First posted 2002-03-25 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-12

CONDITIONS: Chronic Active Epstein-Barr Virus
Keywords: Herpes; Hemophagocytosis; Epstein-Barr Virus; Lymphoproliferative Disease; Mononucleosis; Natural History; Epstein-Barr; EBV; CAEBV; Chronic Active Epstein-Barr Virus; Virus
MeSH Terms: conditions — Herpes Simplex; Epstein-Barr Virus Infections; Lymphoproliferative Disorders; Infectious Mononucleosis; Virus Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAEBV: Patients with chronic active Epstein-Barr virus.
- Hydroa vaccineforme: Patients with EBV hydro vaccineforme.

SUMMARY:
Epstein-Barr virus (EBV) is a member of the human herpes virus family that infects more than 95 percent of the U.S. population. Most infections occur in childhood and cause no symptoms; in adolescents and adults, EBV often causes infectious mononucleosis. It has also been associated with certain forms of cancer. Chronic Epstein-Barr virus (CAEBV) is a rare disease, primarily of children and young adults, that leads to life-threatening infections.

This study seeks to identify genetic mutations responsible for CAEBV. A secondary goal is to learn more about the natural history of CAEBV.

The study will examine blood and tissue samples from up to 50 patients (age 3 and above) with CAEBV and up to 150 of their relatives (age 1 and above). Autopsy samples may be included in the study. Up to 300 anonymous blood samples from the NIH Clinical Center Blood Transfusion Medicine will also be examined for comparison.

No more than 450 milligrams (30 tablespoons) of blood per 8 weeks will be drawn from adult patients, and no more than 7 milliliters per kilogram of blood per 8 weeks will be drawn from patients under age 18. Local health care providers will refer patients to the study and will obtain the samples. Some patients may also be seen at the NIH Clinical Center. Those patients will have a full medical history and physical examination, along with chest X-ray, blood counts, blood chemistry, EBV serologies, and viral load. Other tests, such as CT scan or MRI, may be performed if medically indicated. Patients will be asked to undergo leukapheresis.

In vitro tests on the blood or tissue samples will include analysis for proteins or genes that are involved in the immune response; cloning of portions of patient DNA; transformation of B cells with EBV; measurement of the ability of patient blood cells to kill EBV-infected cells; determination of lymphocyte subsets; and determination of antibodies to EBV or other herpes viruses.

If a genetic cause for CAEBV is found, the investigators will be available to discuss the results with patients in person or by telephone. Genetic indications of risk for other diseases will also be discussed with patients.

...

DETAILED DESCRIPTION:
Patients with chronic active Epstein-Barr virus (CAEBV) have (a) an illness that began as a primary infection with EBV or markedly elevated titers of antibodies to EBV, (b) histological evidence of organ disease, and (c) elevated EBV DNA levels in the blood or EBV DNA or proteins in affected tissues. This is primarily a disease of children and young adults. Many of these patients develop hypogammaglobulinemia or pancytopenia and death is frequently due to opportunistic infections or T cell lymphoproliferative disease. The primary goal of this study is to identify genetic mutations responsible for CAEBV. The secondary goal of this study is to learn more about the natural history of CAEBV. Blood samples or available tissues (e.g., previous biopsy or autopsy material) from patients with CAEBV and their relatives will be analyzed to identify disease genes that are mutated in this population. In addition, some of the patients will be invited to come for evaluation at the NIH Clinical Center. At that time, medically indicated studies of disease progression will be performed. Serial virologic and immunologic studies will be performed. Eligible relatives of patients will be studied to compare the gene(s) associated with CAEBV in patients with the gene(s) in their relatives. Knowledge gained from this study has the potential of providing insights into the immunologic control of EBV infections. In addition, identification of the molecular mechanisms for CAEBV may provide insights leading to improved treatments for this disease.

ELIGIBILITY:
* ELIGIBILITY CRITERIA

CAEBV PATIENTS

Study size: up to 150 patients

Sex distribution: male and female

Age range: 1 year old and above

Patients with known or suspected CAEBV and their relatives will be recruited by referrals from health care providers. The rarity of this disease will markedly limit the number of patients available to study; therefore, we will enroll patients who are 1 year of age and older. However, children under the age of 3 years old will be enrolled as samples- only participants and not be evaluated at the Clinical Center.

Patient recruitment is irrespective of racial and ethnic group or sex. NIAID investigators will be available to answer questions and discuss general aspects of CAEBV and identified genes or modifier genes with participants or their providers.

Eligibility criteria: To be considered having CAEBV, a patient must have:

1. a severe progressive illness that began as a primary EBV infection, or associated with positive EBV-specific antibody titers (IgG-VCA, ; EA or EBNA) not otherwise explained AND
2. evidence of major organ involvement such as lymphadenitis, hemophagocytosis, meningoencephalitis, persistent hepatitis, splenomegaly, interstitial pneumonitis, bone marrow hypoplasia, uveitis AND
3. detection of elevated levels of EBV DNA, RNA or proteins in affected tissues OR elevated levels of EBV DNA in the peripheral blood

Exclusion Criteria:

(a) Any other condition that, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the patient participating in the study.

RELATIVES OF CAEBV PATIENTS:

Study size: up to 150 relatives of CAEBV patients

Age range: 3 years and above

To determine the genetic basis for this syndrome, the evaluation of blood, saliva and/or previously obtained tissue specimens from healthy relatives of CAEBV patients will serve as controls. No tissue biopsies will be performed on healthy relatives. We will

perform some of the studies listed on samples from normal relatives.

UNRELATED VOLUNTEERS

Study size: up to 300 persons

Age range: 18 years and above

Panels of anonymous blood samples will be obtained through NIH Clinical Center Blood Transfusion Medicine to determine if identified genetic changes are mutations or polymorphisms.

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with known or suspected CAEBV and their relatives will be recruited by referrals from health care providers or self-referrals.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2002-04-16 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to identify genetic mutations responsible for CAEBV. | ongoing
  Provide insights into the immunologic control of EBV infections.

SECONDARY OUTCOMES:
The secondary goal of this study is to learn more about the natural history of CAEBV, to assess the viral burden and localization, and to determine if defects are present in pathways involved in cytotoxic functions of T or NK cells. | ongoing
  Identification of the molecular mechanisms fro CAEBV.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Cohen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Okamura T, Hatsukawa Y, Arai H, Inoue M, Kawa K. Blood stem-cell transplantation for chronic active Epstein-Barr virus with lymphoproliferation. Lancet. 2000 Jul 15;356(9225):223-4. doi: 10.1016/S0140-6736(00)02488-0. PMID 10963205
- [Background] Cohen JI, Jaffe ES, Dale JK, Pittaluga S, Heslop HE, Rooney CM, Gottschalk S, Bollard CM, Rao VK, Marques A, Burbelo PD, Turk SP, Fulton R, Wayne AS, Little RF, Cairo MS, El-Mallawany NK, Fowler D, Sportes C, Bishop MR, Wilson W, Straus SE. Characterization and treatment of chronic active Epstein-Barr virus disease: a 28-year experience in the United States. Blood. 2011 Jun 2;117(22):5835-49. doi: 10.1182/blood-2010-11-316745. Epub 2011 Mar 31. PMID 21454450
- [Background] Cohen JI. Optimal treatment for chronic active Epstein-Barr virus disease. Pediatr Transplant. 2009 Jun;13(4):393-6. doi: 10.1111/j.1399-3046.2008.01095.x. No abstract available. PMID 19032417
- [Derived] Cohen JI, Manoli I, Dowdell K, Krogmann TA, Tamura D, Radecki P, Bu W, Turk SP, Liepshutz K, Hornung RL, Fassihi H, Sarkany RP, Bonnycastle LL, Chines PS, Swift AJ, Myers TG, Levoska MA, DiGiovanna JJ, Collins FS, Kraemer KH, Pittaluga S, Jaffe ES. Hydroa vacciniforme-like lymphoproliferative disorder: an EBV disease with a low risk of systemic illness in whites. Blood. 2019 Jun 27;133(26):2753-2764. doi: 10.1182/blood.2018893750. Epub 2019 May 7. PMID 31064750
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-I-0147.html